CLINICAL TRIAL: NCT01720953
Title: Neuropsychiatric Mechanisms of Change in Mentalization Based Treatment of Borderline Personality Disorder (MENTAB)
Acronym: MENTAB
Status: Terminated | Type: Observational
Sponsor: Rune Andersen (Other)
Collaborators: Psychiatry Roskilde (Industry); University of Copenhagen (Other); Psychiatric Epigenetics Laboratory, Institute of Psychiatry, UK (Unknown); University of Southern Denmark (Other); Psychoanalysis Unit, University College London, UK (Unknown); Aarhus University Hospital (Other); University College Zealand, Denmark (Unknown); Research Division of Clinical Biochemistry, Koege Hospital, Denmark (Unknown)
Responsible Party: Sponsor-Investigator, Rune Andersen, Senior researcher, Ph.D., Region Sjælland
Organization: Region Sjælland (Other)
Other Study IDs: SJ-311
Record Dates: First submitted 2012-10-26; First posted 2012-11-02 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2014-07

CONDITIONS: Borderline Personality Disorder
Keywords: Borderline Personality Disorder; Mentalization Based Therapy; DNA methylation; BDNF; Cortisol; Neuropsychology
MeSH Terms: conditions — Borderline Personality Disorder | interventions — Mentalization-Based Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples to measure DNA methylation and BDNF serum levels. Salivary samples to measure cortisol levels.

GROUPS / COHORTS (1):
- Healthy control subjects: Matched healthy control subjects will be assessed at 6 month intervals to compare changes in DNA methylation, BDNF serum levels, salivary cortisol levels, and neuropsychological test performance. Healthy control subjects will within the 1-year study period also undergo continuous assessment for comparative changes in symptoms of dissociation, depression, and personality dysfunction.
  Interventions: Other: Mentalization Based Therapy

INTERVENTIONS:
Other: Mentalization Based Therapy — Fifty female patients diagnosed with BPD will undergo a year of intensive Mentalization Based Therapy that is designed to target domains of BPD pathology. The patients will be assessed at baseline and every 6 months over the treatment period.

SUMMARY:
Purpose:

Borderline personality disorder (BPD) is a complex psychiatric disease of uncertain aetiology and pathogenesis. A key mechanism of disease susceptibility and treatment response could be epigenetic changes in DNA methylation patterns. However, no study has yet demonstrated that psychotherapy can exert its therapeutic effect through epigenetic mechanisms. The main aim of this study is to analyze the promoter methylation pattern of genes considered to be related to the development and psychopathology of BPD, in particular the brain-derived neurotrophic factor (BDNF) and glucocorticoid receptor genes, and the effects of mentalization based treatment (MBT) on changes. Associations to changes in BDNF serum levels and salivary cortisol levels, as well as key components of BPD aetiology and core treatment targets in MBT, will also be investigated. Should epigenetic mechanisms have importance for BPD pathology and effects of treatment, there is potential use of DNA methylation patterns as valid biomarker measures of diagnosis, prognosis, and treatment response.

Hypothesis:

The formation and maintenance of symptoms in BPD is mediated through neuropsychiatric mechanisms that can be affected through psychological treatment. Specifically, aberrant epigenetic regulation of neuropsychiatric genes related to behavioural control and affect regulation, as well as BDNF and cortisol levels, is ameliorated by therapeutic processes.

Method:

Fifty female patients diagnosed with BPD will undergo a year of intensive MBT that is designed to target domains of BPD pathology. The patients will be assessed at baseline and every 6 months over the treatment period. Matched healthy control subjects will be assessed at 6 month intervals to compare changes in DNA methylation, BDNF serum levels, salivary cortisol levels, and neuropsychological test performance. To link components of the neuropsychiatric mechanisms underlying the onset of illness, course, and response to treatment, patients will undergo assessment of clinical symptoms, comorbidity patterns and psychosocial impairment. Patients and control subjects will at baseline undergo assessment for childhood trauma, self-harm, suicidal behavior, early maladaptive schemas, and personality traits, and within the 1-year study period also undergo continuous assessment for changes in symptoms of dissociation, depression, and personality dysfunction.

ELIGIBILITY:
Patients:

Inclusion Criteria:

* Female patients between the ages 18 - 40 with a clinical diagnosis of Borderline Personality Disorder to undergo a year of Mentalization Based Therapy at the Psychiatric Clinic Roskilde.

Exclusion Criteria:

* Severe comorbidity
* Serious medical condition
* Pregnancy

Healthy control subjects:

Inclusion Criteria:

* Match patients on age, gender, and socioeconomic status.

Exclusion Criteria:

* Any mental disorder
* Serious medical condition
* Pregnancy

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Fifty female patients diagnosed with BPD, who will undergo a year of intensive Mentalization Based Therapy at the Psychiatric Clinic Roskilde, Denmark, and a matched healthy control subjects matched on age, gender and socioeconomic status.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-10; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Promoter methylation pattern of genes considered to be related to the development and pathology of BPD, in particular the BDNF and glucocorticoid receptor genes | Assessed at baseline, and after 6 and 12 months
BDNF serum levels | Assessed at baseline, and after 6 and 12 months
Salivary cortisol levels | Assessed at baseline, and after 6 and 12 months
Neuropsychological test performance | Assessed at baseline and after 12 months
  Assessed by a comprehensive battery of neuropsychological tests to measure both cognitive and emotion processing, including standard paper-and-pencil tests (WAIS-IV) and selected computerized tests (CANTAB, SuperLab and E-Prime). An interview will be conducted to assess autobiographical memory function.
Psychopathology | Assessed before baseline, and after 6 and 12 months
  Measured by Zanarini Rating Scale for Borderline Personality Disorder (ZAN-BPD), Hamilton Rating Scale for Depression (HAM-D), Symptom Checklist-90-Revised (SCL-90-R), Severity Indices of Personality Problems (SIPP-118), and Dissociative Experiences Scale - Brief (DES-B)
Affect regulation | Assessed at baseline, and after 6 and 12 months
  Measured by Affective Lability Scale (ALS-18), Barratt Impulsiveness Scale (BIS-11), Buss-Perry Aggression Questionnaire (BPAQ), Toronto Alexithymia Scale (TAS-20)

CONTACTS AND LOCATIONS:
Overall Officials: Erik Simonsen, Professor, MD, Ph.D., Principal Investigator — Psychiatric Research Unit, Region Zealand, Denmark; Rune Andersen, Ph.D., Study Chair — Psychiatric Research Unit, Region Zealand, Denmark
Locations (1):
- Psychiatric Research Unit, Region Zeland, Roskilde, Denmark